CLINICAL TRIAL: NCT03229993
Title: The Safety and Efficacy of OCT in the Evaluation and Treatment of Angiographically Borderline Coronary Artery Lesions
Brief Title: OCT in Borderline Coronary Artery Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCT-20170723
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Optical Coherence Tomography (OCT); Percutaneous Coronary Intervention (PCI); Single-Photon Emission Computed Tomography (SPECT); Coronary Angiography (CAG); Borderline Coronary Artery Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OCT guided PCI (Experimental)
  Interventions: Diagnostic Test: OCT
- OCT guided medicine (Experimental)
  Interventions: Diagnostic Test: OCT
- SPECT guided PCI (No Intervention)
- SPECT guided medicine (No Intervention)

INTERVENTIONS:
Diagnostic Test: OCT — OCT is used to assess whether PCI will be of benefit to the treatment of the borderline coronary artery lesions
  Arms: OCT guided PCI; OCT guided medicine

SUMMARY:
To find out the safety and efficacy of Optical Coherence Tomography (OCT) in the evaluation and treatment of angiographically borderline coronary artery lesions in a Chinese population, and to compare the effectiveness of OCT versus SPECT in treating such subjects. All the participants included in the study will be those that are found to have borderline coronary artery lesions on coronary angiography, in whom the investigators feel that OCT will be useful to assess whether PCI will be of benefit to the treatment of the lesion pathology, or whether optimal medical therapy is the most appropriate treatment modality. Those participants who declined OCT will be offered SPECT as an alternative method to assess and treat the borderline coronary artery stenosis.

It is estimated that OCT guided "PCI or not" has a non-inferiority to SPECT's in the borderline coronary artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study will be only those participants in whom diagnostic coronary angiography revealed borderline coronary artery lesion. These participants will undergo the OCT procedure, or alternatively ECT.

Exclusion Criteria:

* Exclusion criteria will be those participants with previous cardiogenic shock, stroke, renal dysfunction, and acute or chronic total occlusion coronary lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
MACEs | 12 months
  The incidence of major adverse cardiac events (MACEs) including death, myocardial infarction, and stent thrombosis.
TLR | 12 months
  The incidence of target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Rehospitalization | 12 months
  The incidence of rehospitalization due to cardiac events
Recurrent angina | 12 months
  The incidence of recurrent angina

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided